CLINICAL TRIAL: NCT06232265
Title: An Observational Study on Predicting the Efficacy of Immunotherapy for Non-small-cell Lung Cancer Based on LIRAscore
Brief Title: An Observational Study on Predicting the Efficacy of Immunotherapy for NSCLC Based on LIRAscore
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-412
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: immunotherapy; LIRA score; biomarker
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-center, observational clinical study to explore the role of LIRAscore in predicting immunotherapy monotherapy and combination with chemotherapy efficacy and prognosis in locally advanced or metastatic non-small-cell lung cancer. The study plans to enroll 108 patients. The primary endpoint of this study was ORR, and secondary endpoints were PFS, OS, DoR, DCR, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participated in the study, signed the informed consent, and had good compliance;
2. Histologically and/or cytologically confirmed previously untreated, locally advanced or metastatic non-small-cell lung cancer (stage IIIB/IIIC or stage IV) without driver gene mutation;
3. Patients are willing to receive immunotherapy monotherapy or immunotherapy combined with chemotherapy;
4. The patient agrees to provide the remaining tissue samples after clinical routine diagnosis during the baseline period for LIRA score and PD-L1 immunohistochemical testing;
5. The Eastern Organization for Oncology (ECOG) physical fitness score is 0 or 1;
6. The patient has at least one measurable or unmeasurable but evaluable lesion.

Exclusion Criteria:

1. According to clinical routine, patients do not meet the criteria for receiving standard anti-tumor treatment;
2. Patients with known EGFR mutations, ALK rearrangements or ROS1 rearrangements are not eligible to participate in this study;
3. According to the researcher's judgment, the patient is not suitable to participate in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects of this study were patients with previously untreated, locally advanced or metastatic non-small-cell lung cancer (stage IIIB/IIIC or stage IV) without driver gene mutation.
Sampling Method: Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 3 years
  Defined as the proportion of patients who achieved complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | 3 years
  Defined as the time from first recieving treatment to the first occurrence of disease progression or death from any cause determined by IRC based on the Solid Tumor Efficacy Evaluation Criteria (RECIST) 1.1, whichever occurs first
Overall Survival (OS) | 3 years
  Defined as the time from first treatment to death for any reason.
Duration of response (DoR) | 3 years
  Defined as the time from the first recorded objective remission to the disease progression determined by IRC according to RECIST version 1.1, or the time of death from any cause, whichever occurs first.
Disease Control Rate (DCR) | 3 years
  Defined as the proportion of patients whose best overall efficacy (BOR) determined by IRC according to RECIST 1.1 is complete remission, partial remission, or disease stability

CONTACTS AND LOCATIONS:
Overall Officials: Wangjun Liao, MD, PhD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China